CLINICAL TRIAL: NCT04481789
Title: Clinical Pharmacology Study of Oral Edaravone in Healthy Adult Males (Drug Interaction Study and Preliminary Regimen-Finding Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MT-1186-J02
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone; Rosuvastatin Calcium; Sildenafil Citrate; Furosemide

STUDY DESIGN:
Intervention Model Description: Cohort 1 is open-label, non-randomized, sequential, and add-on study. Cohort 2 is single-dose, open-label, randomized, and cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin, Sildenafil, and MT-1186 (Experimental): Group 1 of Cohort 1:
  A single-sequence study in which healthy male subjects receive a single dose of rosuvastatin on Day 1 followed by a single dose of sildenafil on Day 4. MT-1186 will be administered from Day 6 to 13 with co-administration of rosuvastatin and sildenafil on Day 9 and 12, respectively.
  Interventions: Drug: MT-1186; Drug: Rosuvastatin; Drug: Sildenafil
- Furosemide and MT-1186 (Experimental): Group 2 of Cohort 1:
  A single-sequence study in which healthy male subjects receive a single dose of furosemide on Day 1. MT-1186 will be administered from Day 3 to 7 with co-administration of furosemide on Day 6.
  Interventions: Drug: MT-1186; Drug: Furosemide
- MT-1186 (Experimental): Cohort 2:
  A three-way crossover study in which Japanese healthy male subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 4, and 7 according to their treatment sequence with 3-day wash out between doses. Caucasian healthy male subjects receive a single dose of MT-1186 at the same period with Japanese subjects under the corresponding condition on Day 1, 4, or 7 according to their treatment schedule.
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — Suspension
  Other Names: Edaravone
Drug: Rosuvastatin — Tablets
  Other Names: Crestor
  Arms: Rosuvastatin, Sildenafil, and MT-1186
Drug: Sildenafil — Tablets
  Other Names: Viagra
  Arms: Rosuvastatin, Sildenafil, and MT-1186
Drug: Furosemide — Tablets
  Other Names: Lasix
  Arms: Furosemide and MT-1186

SUMMARY:
* Cohort 1: To evaluate the drug interactions, safety, and tolerability of oral edaravone when coadministered with rosuvastatin, sildenafil or furosemide in healthy adult males
* Cohort 2: To evaluate the pharmacokinetics, safety, and tolerability of oral edaravone in healthy Japanese and Caucasian adult males

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteers
* Cohort 1: Japanese, Cohort 2: Japanese or Caucasian
* Subjects aged between 20 and 45 years at the time of informed consent
* Subjects who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects with a current or previous history of cardiac, hepatic, renal, gastrointestinal, respiratory, psychiatric/nervous, hematopoietic, or endocrine diseases, and those whom the investigator (or subinvestigator) deems unsuitable for the study
* Body mass index (BMI) of <18.0 or >30.0, or body weight of <50 kg (BMI formula: body weight [kg]/height [m]2, rounded to one decimal place)
* Subjects who have undergone any surgery known to affect the gastrointestinal absorption of drugs
* Subjects who do not agree to use an effective method of contraception from initiation of study drug administration to 14 days after completion (discontinuation) of study drug administration
* Subjects who have previously received edaravone
* Subjects who have participated in another clinical study and received a study drug within 12 weeks before providing informed consent
* Use of any drug(s) other than the study drug or as-needed use of acetylsalicylic acid within 7 days before the initiation of study drug or victim drug administration
* Use of any alcohol, xanthine, or caffeine-containing product(s) within 24 hours before screening and Day -1 visiting
* Use of any supplement(s) within 7 days before the initiation of study drug or victim drug administration
* Use of grapefruit, grapefruit juice, or any processed food(s) containing these substances during the following periods (Cohort 1: within 7 days before the initiation of victim drug administration, Cohort 2: within 24 hours before each Day -1 visiting)
* Use of any tobacco or nicotine-containing product(s) (Cohort 1: within 12 weeks before the initiation of victim drug administration during the following periods, Cohort 2: within 24 hours before each Day -1 visiting)
* Use of any health food(s) containing St John's Wort (Hypericum perforatum) within 2 weeks before the initiation of victim drug administration (only in Cohort 1)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shimizu H, Nishimura Y, Shiide Y, Akimoto M, Matsuda H, Kato Y, Hirai M. Food Effect Study to Assess the Impact on Edaravone Pharmacokinetic Profiles in Healthy Participants. Clin Ther. 2022 Dec;44(12):1552-1565. doi: 10.1016/j.clinthera.2022.10.001. Epub 2022 Nov 12. PMID 36376130
- [Result] Shimizu H, Nishimura Y, Shiide Y, Matsuda H, Akimoto M, Matsuda M, Nakamaru Y, Kato Y, Kondo K. Evaluation of Pharmacokinetics, Safety, and Drug-Drug Interactions of an Oral Suspension of Edaravone in Healthy Adults. Clin Pharmacol Drug Dev. 2021 Oct;10(10):1174-1187. doi: 10.1002/cpdd.925. Epub 2021 Mar 11. PMID 33704925

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1: A single-sequence study in which healthy male subjects receive a single dose of rosuvastatin on Day 1 followed by a single dose of sildenafil on Day 4. Oral edaravone will be administered from Day 6 to 13 with co-administration of rosuvastatin and sildenafil on Day 9 and 12, respectively.
- Furosemide and Edaravone Group 2 of Cohort 1: A single-sequence study in which healthy male subjects receive a single dose of furosemide on Day 1. Oral edaravone will be administered from Day 3 to 7 with co-administration of furosemide on Day 6.
- Edaravone Group 3 of Cohort 2: A three-way crossover study in which Japanese healthy male subjects receive a single dose of Oral edaravone under several dosing condition on Day 1, 4, and 7 according to their treatment sequence with 3-day wash out between doses.
  Period 1:Japanese subjects receive a single dose of Edaravone under fasted condition on Day 1.
  Period 2: Japanese subjects receive a single dose of Edaravone1 hour before a high-fat meal on Day 4.
  Period 3: Japanese subjects receive a single dose of Edaravone 4 hours after a high-fat meal on Day 7.
- Edaravone Group 4 of Cohort 2: A three-way crossover study in which Japanese healthy male subjects receive a single dose of Oral edaravone under several dosing condition on Day 1, 4, and 7 according to their treatment sequence with 3-day wash out between doses.
  Period 1: Japanese subjects receive a single dose of Edaravone 4 hours after a high-fat meal.
  Period 2: Japanese subjects receive a single dose of Edaravone under fasted condition.
  Period 3: Japanese subjects receive a single dose of Edaravone1 hour before a high-fat meal.
- Edaravone Group 5 of Cohort 2: A three-way crossover study in which Japanese healthy male subjects receive a single dose o Oral edaravone under several dosing condition on Day 1, 4, and 7 according to their treatment sequence with 3-day wash out between doses.
  Period 1: Japanese subjects receive a single dose of Edaravone1 hour before a high-fat meal.
  Period 2: Japanese subjects receive a single dose of Edaravone 4 hours after a high-fat meal.
  Period 3: Japanese subjects receive a single dose of Edaravone under fasted condition.
- Caucasian Group of Cohort 2: Caucasian healthy male subjects receive a single dose of MT-1186 under fasted condition at the same period with Japanese subjects on Day 1, 4, or 7 according to their treatment schedule.
Period: Period 1
Arm/Group | Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1 | Furosemide and Edaravone Group 2 of Cohort 1 | Edaravone Group 3 of Cohort 2 | Edaravone Group 4 of Cohort 2 | Edaravone Group 5 of Cohort 2 | Caucasian Group of Cohort 2
Started | 32 | 34 | 3 | 3 | 3 | 3
Completed | 31 | 34 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1 | Furosemide and Edaravone Group 2 of Cohort 1 | Edaravone Group 3 of Cohort 2 | Edaravone Group 4 of Cohort 2 | Edaravone Group 5 of Cohort 2 | Caucasian Group of Cohort 2
Started | 31 | 34 | 3 | 3 | 3 | 3
Completed | 31 | 34 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1 | Furosemide and Edaravone Group 2 of Cohort 1 | Edaravone Group 3 of Cohort 2 | Edaravone Group 4 of Cohort 2 | Edaravone Group 5 of Cohort 2 | Caucasian Group of Cohort 2
Started | 31 | 0 (Cohort 1 Group 2 was planned as a 2-period study. Therefore, Period 3 was not conducted.) | 3 | 3 | 3 | 3
Completed | 31 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1: A single-sequence study in which healthy male subjects receive a single dose of rosuvastatin on Day 1 followed by a single dose of sildenafil on Day 4. MT-1186 will be administered from Day 6 to 13 with co-administration of rosuvastatin and sildenafil on Day 9 and 12, respectively.
- Furosemide and Edaravone Group 2 of Cohort 1: A single-sequence study in which healthy male subjects receive a single dose of furosemide on Day 1. MT-1186 will be administered from Day 3 to 7 with co-administration of furosemide on Day 6.
- Japanese Combined of Cohort 2: A three-way crossover study in which Japanese healthy male subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 4, and 7 according to their treatment sequence with 3-day wash out between doses.
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin, Sildenafil, and Edaravone Group 1 of Cohort 1 | Furosemide and Edaravone Group 2 of Cohort 1 | Japanese Combined of Cohort 2 | Caucasian Group of Cohort 2 | Total
Number analyzed (Participants) | 32 | 34 | 9 | 9 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 9 | 9 | 84
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 32 | 34 | 9 | 9 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 32 | 34 | 9 | 0 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 9 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Rosuvastatin, Sildenafil and Furosemide.
Time Frame: Before rosuvastatin dosing and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hrs post-dose, Before sildenafil dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hrs post-dose, Before furosemide dosing and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hrs post-dose
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone.
  DDI effects of oral edaravone was evaluated based on the number of subjects in each period in Cohort 1 (Group 1: Period 1 to 3, Group 2: Period 1 and 2).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Rosuvastatin Alone: Group 1 of Cohort 1: The subjects receive a single dose of rosuvastatin on Day 1.
- Rosubastatin + Edaravone: Group 1 of Cohort 1: The subjects receive edaravone from Day 6 to 13 with co-administration of rosuvastatin on Day 9.
- Sildenafil Alone: Group 1 of Cohort 1: The subjects receive a single dose of sildenafil on Day 4.
- Sildenafil + Edaravone: Group 1 of Cohort 1: The subjects receive edaravone from Day 6 to 13 with co-administration of sildenafil on Day 12.
- Furosemide Alone: Group 2 of Cohort 1: The subjects receive a single dose of furosemide on Day 1.
- Furosemide + Edaravone: Group 2 of Cohort 1: The subjects receive edaravone from Day 3 to 7 with co-administration of furosemide on Day 6.
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Rosubastatin + Edaravone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Sildenafil + Edaravone: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Furosemide + Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 32 | 31 | 31 | 31 | 34 | 34
ng*h/mL | 161 (66.8) | 165 (60.2) | 532 (236) | 482 (195) | 3861 (1031) | 3906 (736.2)
Statistical Analysis 1: Comparison: Rosuvastatin Alone: Group 1 of Cohort 1 vs Rosubastatin + Edaravone: Group 1 of Cohort 1; PK parameters of rosuvastatin, sildenafil, and furosemide alone and in the presence of edaravone were analyzed for the assessments of effect on PK of rosuvastatin, sildenafil, and furosemide by edaravone; Test type: Other — Estimates of least squares mean difference of log-transformed PK parameters between treatments were obtained with their 2-sided 90%CIs for the difference. These estimates and limits were then back-transformed to obtain ratios of least squares geometric means. If the 90%CIs lay entirely within the limits of 0.80 to 1.25, this would provide evidence of no effect of edaravone on the PK of rosuvastatin, sildenafil, and furosemide (LS Mean Ratio: Rosuvastatin + Edaravone / Rosuvastatin Alone); LS Mean Ratio = 1.02, 90% CI 2-sided [0.97 to 1.08]
Statistical Analysis 2: Comparison: Sildenafil Alone: Group 1 of Cohort 1 vs Sildenafil + Edaravone: Group 1 of Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Other — Estimates of least squares mean difference of log-transformed PK parameters between treatments were obtained with their 2-sided 90%CIs for the difference. These estimates and limits were then back-transformed to obtain ratios of least squares geometric means. If the 90%CIs lay entirely within the limits of 0.80 to 1.25, this would provide evidence of no effect of edaravone on the PK of rosuvastatin, sildenafil, and furosemide (LS Mean Ratio: Sildenafil + Edaravone / Sildenafil Alone); LS Mean Ratio = 0.93, 90% CI 2-sided [0.88 to 0.99]
Statistical Analysis 3: Comparison: Furosemide Alone: Group 2 of Cohort 1 vs Furosemide + Edaravone: Group 2 of Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Other — Estimates of least squares mean difference of log-transformed PK parameters between treatments were obtained with their 2-sided 90%CIs for the difference. These estimates and limits were then back-transformed to obtain ratios of least squares geometric means. If the 90%CIs lay entirely within the limits of 0.80 to 1.25, this would provide evidence of no effect of edaravone on the PK of rosuvastatin, sildenafil, and furosemide (LS Mean Ratio: Furosemide + Edaravone / Furosemide Alone); LS Mean Ratio = 1.03, 90% CI 2-sided [0.98 to 1.09]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Rosuvastatin, Sildenafil and Furosemide.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Rosubastatin + Edaravone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Sildenafil + Edaravone: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Furosemide + Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 32 | 31 | 31 | 31 | 34 | 34
ng/mL | 11.3 (5.0) | 11.3 (5.0) | 232 (135) | 201 (97.9) | 1676 (777.7) | 1701 (506.5)
Statistical Analysis 1: Comparison: Rosuvastatin Alone: Group 1 of Cohort 1 vs Rosubastatin + Edaravone: Group 1 of Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Other — Estimates of least squares mean difference of log-transformed PK parameters between treatments were obtained with their 2-sided 90%CIs for the difference. These estimates and limits were then back-transformed to obtain ratios of least squares geometric means. If the 90%CIs lay entirely within the limits of 0.80 to 1.25, this would provide evidence of no effect of edaravone on the PK of rosuvastatin, sildenafil, and furosemide (LS Mean Ratio: Rosuvastatin + Edaravone / Rosuvastatin); LS Mean Ratio = 0.98, 90% CI 2-sided [0.91 to 1.06]
Statistical Analysis 2: Comparison: Sildenafil Alone: Group 1 of Cohort 1 vs Sildenafil + Edaravone: Group 1 of Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; LS Mean Ratio = 0.94, 90% CI 2-sided [0.80 to 1.10]
Statistical Analysis 3: Comparison: Furosemide Alone: Group 2 of Cohort 1 vs Furosemide + Edaravone: Group 2 of Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; LS Mean Ratio = 1.08, 90% CI 2-sided [0.96 to 1.23]

3. Primary Outcome: Tmax of Rosuvastatin, Sildenafil and Furosemide.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Rosubastatin + Edaravone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Sildenafil + Edaravone: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Furosemide + Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 32 | 31 | 31 | 31 | 34 | 34
h | 4.6 (1.5) | 5.1 (1.4) | 0.8 (0.4) | 0.9 (0.5) | 1.7 (1.1) | 1.8 (1.1)

4. Primary Outcome: T1/2 of Rosuvastatin, Sildenafil and Furosemide.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Rosubastatin + Edaravone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Sildenafil + Edaravone: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Furosemide + Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 32 | 31 | 31 | 31 | 34 | 34
h | 14.4 (4.0) | 12.1 (2.2) | 2.8 (1.1) | 3.5 (1.4) | 6.9 (3.5) | 5.8 (3.8)

5. Primary Outcome: AUC0-inf of Unchanged Edaravone.
Time Frame: Group 1 (Day 6, 9 and 12) and Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone. DDI effects of oral edaravone was evaluated based on the number of subjects in each period in Cohort 1 (Group 1: Period 1 to 3, Group 2: Period 1 and 2). Day 3 of Group 1 and Day 9 and 12 of Group 2 were zero participant because no data was collected.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Rosuvastatin, Sildenafil, and Edaravone: Group 1 of Cohort 1: Edaravone was administered once daily for 8 days from Day 6 to 13 with coadministration of rosuvastatin ond Day 9 and sildenafil on Day 12
- Furosemide and Edaravone: Group 2 of Cohort 1: Edaravone was administered once daily for 5 days from Day 3 to 7 with coadministration of furosemide on Day 6.
Arm/Group | Rosuvastatin, Sildenafil, and Edaravone: Group 1 of Cohort 1 | Furosemide and Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 31 | 34
ng*h/mL
  Day 3: Group 2 (Edaravone alone): number analyzed (Participants) | 0 | 34
  Day 3: Group 2 (Edaravone alone) |  | 2535 (919)
  Day 6: Group 1 (Edaravpne alone), Group 2 (Edaravone + Furosemide) | 2616 (730) | 2746 (1015)
  Day 9: Group 1 (Edaravone + Rosuvastatin), Group 2 Not Applicable: number analyzed (Participants) | 31 | 0
  Day 9: Group 1 (Edaravone + Rosuvastatin), Group 2 Not Applicable | 2591 (671) |
  Day 12: Group 1 (Edaravone + Sildenafil), Group 2 Not Applicable: number analyzed (Participants) | 31 | 0
  Day 12: Group 1 (Edaravone + Sildenafil), Group 2 Not Applicable | 2656 (712) |

6. Primary Outcome: Cmax of Unchanged Edaravone.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 1 of Cohort 1: Edaravone was administered once daily for 8 days from Day 6 to 13 with coadministration of rosuvastatin ond Day 9 and sildenafil on Day 12
Arm/Group | Group 1 of Cohort 1 | Furosemide and Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 31 | 34
ng/mL
  Day 3: Group 2 (Edaravone alone): number analyzed (Participants) | 0 | 34
  Day 3: Group 2 (Edaravone alone) |  | 2180 (1035)
  Day 6: Group 1 (Edaravpne alone), Group 2 (Edaravone + Furosemide) | 2724 (1533) | 2074 (1051)
  Day 9: Group 1 (Edaravone + Rosuvastatin): number analyzed (Participants) | 31 | 0
  Day 9: Group 1 (Edaravone + Rosuvastatin) | 2302 (943) |
  Day 12: Group 1 (Edaravone + Sildenafil): number analyzed (Participants) | 31 | 0
  Day 12: Group 1 (Edaravone + Sildenafil) | 2455 (1111) |

7. Primary Outcome: Tmax of Unchanged Edaravone.
Time Frame: as for outcome 5
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone.
  DDI effects of oral edaravone was evaluated based on the number of subjects in each period in Cohort 1 (Group 1: Period 1 to 3, Group 2: Period 1 and 2).
  Day 3 of Group 1 and Day 9 and 12 of Group 2 were zero participants because no data was collected.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 1 of Cohort 1 | Furosemide and Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 31 | 34
h
  Day 3: Group 2 (Edaravone alone): number analyzed (Participants) | 0 | 34
  Day 3: Group 2 (Edaravone alone) |  | 0.34 (0.19)
  Day 6: Group 1 (Edaravpne alone), Group 2 (Edaravone + Furosemide) | 0.30 (0.10) | 0.34 (0.17)
  Day 9: Group 1 (Edaravone + Rosuvastatin): number analyzed (Participants) | 31 | 0
  Day 9: Group 1 (Edaravone + Rosuvastatin) | 0.34 (0.13) |
  Day 12: Group 1 (Edaravone + Sildenafil): number analyzed (Participants) | 31 | 0
  Day 12: Group 1 (Edaravone + Sildenafil) | 0.32 (0.17) |

8. Primary Outcome: T1/2 of Unchanged Edaravone.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 1 of Cohort 1 | Furosemide and Edaravone: Group 2 of Cohort 1
Number analyzed (Participants) | 31 | 34
h
  Day 3: Group 2 (Edaravone alone): number analyzed (Participants) | 0 | 34
  Day 3: Group 2 (Edaravone alone) |  | 4.67 (0.92)
  Day 6: Group 1 (Edaravpne alone), Group 2 (Edaravone + Furosemide) | 5.23 (1.11) | 5.52 (0.60)
  Day 9: Group 1 (Edaravone + Rosuvastatin): number analyzed (Participants) | 31 | 0
  Day 9: Group 1 (Edaravone + Rosuvastatin) | 6.60 (1.18) |
  Day 12: Group 1 (Edaravone + Sildenafil): number analyzed (Participants) | 31 | 0
  Day 12: Group 1 (Edaravone + Sildenafil) | 6.69 (1.31) |

9. Primary Outcome: AUC0-inf of Sulfate Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone.
  DDI effects of oral edaravone was evaluated based on the number of subjects in each period in Cohort 1 (Group 1: Period 1 to 3, Group 2: Period 1 and 2). Sulfate and glucuronide conjugates were not measured in Cohort 1 Group 1.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Group 2 of Cohort 1: Edaravone was administered once daily for 5 days from Day 3 to 7 with coadministration of furosemide on Day 6.
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
ng*h/mL
  Day 3: Group 2 (Edaravone alone) | 26576 (6820)
  Day 6: Group 2 (Edaravone + Furosemide) | 30588 (7064)

10. Primary Outcome: Cmax of Sulfate Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
ng/mL
  Day 3: Group 2 (Edaravone alone) | 8115 (1775)
  Day 6: Group 2 (Edaravone + Furosemide) | 8702 (2147)

11. Primary Outcome: Tmax of Sulfate Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
h
  Day 3: Group 2 (Edaravone alone) | 0.76 (0.28)
  Day 6: Group 2 (Edaravone + Furosemide) | 0.81 (0.30)

12. Primary Outcome: T1/2 of Sulfate Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
h
  Day 3: Group 2 (Edaravone alone) | 3.89 (0.25)
  Day 6: Group 2 (Edaravone + Furosemide) | 4.20 (0.33)

13. Primary Outcome: AUC0-inf of Glucuronide Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
ng*h/mL
  Day 3: Group 2 (Edaravone alone) | 4817 (1282)
  Day 6: Group 2 (Edaravone + Furosemide) | 4953 (1285)

14. Primary Outcome: Cmax of Glucuronide Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
ng/mL
  Day 3: Group 2 (Edaravone alone) | 2318 (649)
  Day 6: Group 2 (Edaravone + Furosemide) | 2304 (694)

15. Primary Outcome: Tmax of Glucuronide Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
h
  Day 3: Group 2 (Edaravone alone) | 0.61 (0.26)
  Day 6: Group 2 (Edaravone + Furosemide) | 0.57 (0.18)

16. Primary Outcome: T1/2 of Glucuronide Conjugate.
Time Frame: Group 2 (Day 3 and 6): Pre-dose, 0.083, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group 2 of Cohort 1
Number analyzed (Participants) | 34
h
  Day 3: Group 2 (Edaravone alone) | 3.65 (0.28)
  Day 6: Group 2 (Edaravone + Furosemide) | 3.97 (0.31)

17. Primary Outcome: AUC0-inf of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone. Three groups of randomized Japanese subjects received a single dose of edaravone under each of 3 dosing meal conditions in a 3-way, 3-period crossover fashion (3X3) in Cohort 2.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Edaravone Single Dose Under Fasting Condition; Edaravone Single Dose 1 Hour After a High-fat Meal; Edaravone Single Dose 4 Hours After a High-fat Meal: Japanese combined
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
ng*h/mL | 1647 (433) | 1475 (658) | 1247 (425)
Statistical Analysis 1: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 1 Hour After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — Estimated difference in least squares means and corresponding 90%CI of log-transformed PK parameters were back transformed to obtain the estimate and CI of the geometric mean ratio of 1 Hour After a High-fat Meal condition to the fasted state; LS Mean Ratio = 0.842, 90% CI 2-sided [0.697 to 1.017]
Statistical Analysis 2: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 4 Hours After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — Estimated difference in least squares means and corresponding 90% CI of log-transformed PK parameters were back transformed to obtain the estimate and CI of the geometric mean ratio of 4 Hours After a High-fat Meal condition to the fasted state; LS Mean Ratio = 0.737, 90% CI 2-sided [0.610 to 0.891]

18. Primary Outcome: Cmax of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 1810 (849.8) | 1502 (1272) | 1012 (603.3)
Statistical Analysis 1: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 1 Hour After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — Estimated difference in least squares means and corresponding 90% CI of log-transformed PK parameters were back transformed to obtain the estimate and CI of the geometric mean ratio of 1 Hour After a High-fat Meal condition to the fasted state; LS Mean Ratio = 0.657, 90% CI 2-sided [0.379 to 1.137]
Statistical Analysis 2: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 4 Hours After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — Estimated difference in least squares means and corresponding 90%CI of log-transformed PK parameters were back transformed to obtain the estimate and CI of the geometric mean ratio of 4 Hours After a High-fat Meal condition to the fasted state; LS Mean Ratio = 0.522, 90% CI 2-sided [0.301 to 0.903]

19. Primary Outcome: Tmax of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
h | 0.25 [0.25 to 1.00] | 0.50 [0.25 to 1.50] | 0.25 [0.25 to 1.00]

20. Primary Outcome: T1/2 of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
h | 9.33 (4.87) | 9.65 (5.41) | 7.66 (4.12)

21. Primary Outcome: AUCinf of Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
ng*h/mL
  Sulfate conjugate | 24484 (5861) | 22689 (6334) | 23022 (5094)
  Glucuronide conjugate | 4178 (873) | 4099 (637) | 3557 (879)

22. Primary Outcome: Cmax of Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
ng/mL
  Sulfate conjugate | 8394 (1609) | 7802 (1556) | 8152 (1731)
  Glucuronide conjugate | 2391 (508) | 2176 (475) | 1924 (380)

23. Primary Outcome: Tmax of Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
h
  Sulfate conjugate | 0.67 (0.25) | 0.91 (0.39) | 0.72 (0.26)
  Glucuronide conjugate | 0.53 (0.20) | 0.76 (0.35) | 0.72 (0.26)

24. Primary Outcome: T1/2 of Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 1 Hour After a High-fat Meal | Edaravone Single Dose 4 Hours After a High-fat Meal
Number analyzed (Participants) | 9 | 9 | 9
h
  Sulfate conjugate | 10.50 (7.67) | 7.53 (3.55) | 7.55 (2.47)
  Glucuronide conjugate | 4.26 (0.38) | 3.89 (0.79) | 3.88 (0.55)

25. Primary Outcome: T1/2 of Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Measure: Mean (Standard Deviation); unit: h
Groups:
- Japanese: Japanese: Edaravone single dose under fasting condition
- White: White: Edaravone single dose under fasting condition
Arm/Group | Japanese | White
Number analyzed (Participants) | 9 | 9
h | 4.26 (0.38) | 4.35 (0.25)

26. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Day 1 to 20 in group 1 of cohort 1, Day 1 to 14 in group 2 of cohort 1, Day 1 to 14 of cohort 2
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Groups:
- Rosuvastatin Alone: Group 1 of Cohort 1: Day 1 to Day 4. The subjects receive a single dose of rosuvastatin on Day 1.
- Sildenafil Alone: Group 1 of Cohort 1: Day 4 to Day 5. The subjects receive a single dose of sildenafil on Day 4.
- Edaravone Alone: Group 1 of Cohort 1: Day 6 to Day 8. The subjects receive a single dose of edaravone from Day 6 to Day 8.
- Edaravone + Rosuvastatin: Group 1 of Cohort 1: Day 9 to Day 11. The subjects receive edaravone from Day 6 to 11 with co-administration of rosuvastatin on Day 9.
- Edaravone + Sildenafil: Group 1 of Cohort 1: Day 12 to Day 20 including end of study assessment. The subjects receive edaravone from Day 12 and 13 with co-administration of sildenafil on Day 12.
- Combined: After Day 6: Group 1 of Cohort 1: Day 6 to Day 20 including end of study assessment.
- Furosemide Alone: Group 2 of Cohort 1: Day 1 to Day 2. The subjects receive a single dose of furosemide on Day 1.
- Edaravone Alone: Group 2 of Cohort 1: Day 3 to Day 5. The subjects receive a single dose of edaravone from Day 3 to Day 5.
- Edaravone + Furosemide: Group 2 of Cohort 1: Day 6 to Day 14 including end of study assessment. The subjects receive edaravone on Day 6 to Day 7 with co-administration of furosemide on Day 6.
- Combined : After Day 3: Group 2 of Cohort 1: Day 3 to Day 14 including end of study assessment.
- Edaravone Single Dose Under Fasting Condition: Japanese Conmibed; Edaravone Single Dose 1 Hour After a High-fat Meal: Japanese Conmibed; Edaravone Single Dose 4 Hours After a High-fat Meal: Japanese Conmibed: Japanese combined
- Edaravone Single Dose Under Fasting Condition: White Conbined: White combined
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Edaravone Alone: Group 1 of Cohort 1 | Edaravone + Rosuvastatin: Group 1 of Cohort 1 | Edaravone + Sildenafil: Group 1 of Cohort 1 | Combined: After Day 6: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Edaravone Alone: Group 2 of Cohort 1 | Edaravone + Furosemide: Group 2 of Cohort 1 | Combined : After Day 3: Group 2 of Cohort 1 | Edaravone Single Dose Under Fasting Condition: Japanese Conmibed | Edaravone Single Dose 1 Hour After a High-fat Meal: Japanese Conmibed | Edaravone Single Dose 4 Hours After a High-fat Meal: Japanese Conmibed | Edaravone Single Dose Under Fasting Condition: White Conbined
Number analyzed (Participants) | 32 | 31 | 31 | 31 | 31 | 31 | 34 | 34 | 34 | 34 | 9 | 9 | 9 | 9
Participants
  Number of Participants with Adverse events | 0 | 2 | 0 | 6 | 3 | 8 | 1 | 0 | 7 | 7 | 0 | 2 | 0 | 0
  Number of Participants with adverse drug reactions | 0 | 0 | 0 | 5 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

27. Secondary Outcome: AUCinf of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: This study was conducted in 2 cohorts; the first cohort assessed DDIs with multiple doses of oral edaravone, and the second cohort evaluated PK and racial differences in PK parameters with oral administration of edaravone. 18 subjects (9 Japanese and 9 White) were enrolled in Cohort 2.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Japanese | White
Number analyzed (Participants) | 9 | 9
ng*h/mL
  Unchanged edaravone | 1647 (433) | 1423 (391)
  Sulfate conjugate | 24484 (5861) | 20098 (1592)
  Glucuronide conjugate | 4178 (873) | 3795 (571)

28. Secondary Outcome: Cmax of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese | White
Number analyzed (Participants) | 9 | 9
ng/mL
  Unchanged edaravone | 1810 (850) | 1484 (920)
  Sulfate conjugate | 8394 (1609) | 6530 (787)
  Glucuronide conjugate | 2391 (508) | 2136 (403)

29. Secondary Outcome: Tmax of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Japanese | White
Number analyzed (Participants) | 9 | 9
h
  Unchanged edaravone | 0.4 (0.3) | 0.4 (0.2)
  Sulfate conjugate | 0.67 (0.25) | 0.67 (0.25)
  Glucuronide conjugate | 0.53 (0.20) | 0.61 (0.22)

30. Secondary Outcome: T1/2 of Unchanged Edaravone.
Time Frame: Before dosing, and 0.083, 0.25, 0.5 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Japanese | White
Number analyzed (Participants) | 9 | 9
h
  Unchanged edaravone | 9.3 (4.9) | 16.2 (15.8)
  Sulfate conjugate | 10.5 (7.7) | 10.7 (6.5)
  Glucuronide conjugate | 4.3 (0.4) | 4.4 (0.3)

ADVERSE EVENTS:
Time Frame: Cohort 1 Group 1: Day 1 to Day 20. Cohort 1 Group 2 and Cohort 2: Day 1 to Day 14.
Description: This study was conducted in 2 cohorts; the first cohort assessed DDIs, and the second cohort evaluated PK and racial differences in PK parameters with oral edaravone. DDI effects of oral edaravone was evaluated based on the number of subjects in each period in Cohort 1 (Group 1: Period 1 to 3, Group 2: Period 1 and 2). Three groups of randomized Japanese subjects received a single dose of edaravone under each of 3 dosing meal conditions in a 3-way, 3-period crossover fashion (3X3) in Cohort 2.
Groups:
- Edaravone Single Dose Under Fasting Condition: White Combined: White combined
Arm/Group | Rosuvastatin Alone: Group 1 of Cohort 1 | Sildenafil Alone: Group 1 of Cohort 1 | Edaravone Alone: Group 1 of Cohort 1 | Edaravone + Rosuvastatin: Group 1 of Cohort 1 | Edaravone + Sildenafil: Group 1 of Cohort 1 | Combined: After Day 6: Group 1 of Cohort 1 | Furosemide Alone: Group 2 of Cohort 1 | Edaravone Alone: Group 2 of Cohort 1 | Edaravone + Furosemide: Group 2 of Cohort 1 | Combined : After Day 3: Group 2 of Cohort 1 | Edaravone Single Dose Under Fasting Condition: Japanese Conmibed | Edaravone Single Dose 1 Hour After a High-fat Meal: Japanese Conmibed | Edaravone Single Dose 4 Hours After a High-fat Meal: Japanese Conmibed | Edaravone Single Dose Under Fasting Condition: White Combined
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/34 | 0/34 | 0/34 | 0/34 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/34 | 0/34 | 0/34 | 0/34 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/32 | 2/31 | 0/31 | 6/31 | 3/31 | 8/31 | 1/34 | 0/34 | 7/34 | 7/34 | 0/9 | 2/9 | 0/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin Alone: Group 1 of Cohort 1 (N=32) | Sildenafil Alone: Group 1 of Cohort 1 (N=31) | Edaravone Alone: Group 1 of Cohort 1 (N=31) | Edaravone + Rosuvastatin: Group 1 of Cohort 1 (N=31) | Edaravone + Sildenafil: Group 1 of Cohort 1 (N=31) | Combined: After Day 6: Group 1 of Cohort 1 (N=31) | Furosemide Alone: Group 2 of Cohort 1 (N=34) | Edaravone Alone: Group 2 of Cohort 1 (N=34) | Edaravone + Furosemide: Group 2 of Cohort 1 (N=34) | Combined : After Day 3: Group 2 of Cohort 1 (N=34) | Edaravone Single Dose Under Fasting Condition: Japanese Conmibed (N=9) | Edaravone Single Dose 1 Hour After a High-fat Meal: Japanese Conmibed (N=9) | Edaravone Single Dose 4 Hours After a High-fat Meal: Japanese Conmibed (N=9) | Edaravone Single Dose Under Fasting Condition: White Combined (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04481789/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT04481789/SAP_001.pdf